CLINICAL TRIAL: NCT02596178
Title: Titration of PEEP During Mechanical Ventilation in Patients With ARDS Using Electrical Impedance Tomography.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Research team no longer available.
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Brian Walsh, Co-Investigator, Boston Children's Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-P00017859
Record Dates: First submitted 2015-11-02; First posted 2015-11-04 (Estimated); Last update posted 2019-06-05 (Actual); Status verified 2019-06

CONDITIONS: Acute Respiratory Distress Syndrome
MeSH Terms: conditions — Respiratory Distress Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- EIT Guided PEEP Therapy (Experimental)
  Interventions: Device: Electrical Impedance Tomography

INTERVENTIONS:
Device: Electrical Impedance Tomography — Electrical impedance tomography capitalizes on changes in electrical impendence between air-filled versus tissue or fluid-filled spaces in order to characterize and quantify regional distribution of lung volume at the bedside.

SUMMARY:
Lung units that participate in gas exchange are known as 'recruited' lung. Patients with lung injury suffer from a proportion of units that do not participate in gas exchange (i.e. the derecruited lung), which results in impaired gas exchange and induces an inflammatory cascade. The level of PEEP is often coupled to indices of oxygenation such as PaO2, PaO2 to FIO2 ratio, or oxygen index. Currently, two strategies are widely accepted and considered equivocal, one strategy using a lower PEEP level coupled to a certain oxygen requirement, the other using a higher PEEP level.

The primary purpose of this study is to demonstrate the safety and efficacy of an electrical impedance tomography (EIT) PEEP titration protocol designed to recruit collapsed lung in children with ARDS and properly maintain lung volumes by setting an optimal PEEP level. A safety system has been developed using the ARDSnet FIO2/PEEP High (upper threshold limit) and Low (lower threshold limit) algorithm. Efficacy will be defined as an improvement in lung volume as assessed by electrical impedance tomography, lung compliance and by an improvement in markers of gas exchange. Safety will be defined as the incidence of barotrauma and hemodynamic consequences that occur during the protocol. Those results will be compared to incidences of barotrauma and hemodynamic compromise within the ARDS literature. Knowledge gained from this pilot will be instrumental in developing an EIT imagine guided protocol which will allow us to conduct future RCTs utilizing EIT technology

DETAILED DESCRIPTION:
Currently, clinical practice regarding positive end expiratory pressure (PEEP) strategies for Acute Respiratory Distress Syndrome (ARDS) revolves around two PEEP/FIO2 algorithms developed NHLBI research ARDSnet program. These two algorithms are known as the "High" PEEP/ lower FIO2 and "Low" PEEP/ higher FIO2 protocols. The High PEEP/ lower FIO2 protocol is seen as aggressive or the highest PEEP level a clinician would want to set, while the low PEEP/ higher FIO2 is seen as lowest PEEP level a clinician would set. While many studies have demonstrated safety and efficacy of a PEEP setting based on a required fraction of inspired oxygen (FIO2) to maintain adequate oxygenation, yet there are equal outcomes between the two strategies. There is growing evidence that the Low PEEP/ higher FIO2 protocol leaves large proportions of the lung derecruited and the High PEEP/FIO2 protocol may create overdistension in the compliant sections of the lung that are largely free from disease as it uses a single gas exchange (oxygenation) parameter to determine PEEP settings.

Specific Aim 1: To demonstrate safety of an EIT guided PEEP titration strategy. (Hypothesis: EIT guided titration of PEEP will improve ventilation and oxygenation without increasing incidence of barotrauma or hemodynamic compromise.)

Specific Aim 2: To demonstrate the efficacy of a PEEP titration strategy to increase distribution of ventilation and improve oxygenation in children with ARDS utilizing an EIT guided protocol within two standards of care. (Hypothesis: EIT guided titration of PEEP will lead to a more homogeneous distribution of ventilation, improved lung compliance and improved ventilation and oxygenation.) Background and Significance Lung units participating in gas exchange are known as 'recruited' lung. Patients with lung injury suffer from a proportion of lung units which not participating in gas exchange (i.e. the derecruited state), at times resulting in impaired gas exchange. Derecruitment of alveoli may also cause intrapulmonary shunting and worsen lung injury through atelectotrauma. Outcomes in ARDS have improved significantly since clinicians have begun to employ lung protective strategies, including low-tidal volume ventilation and permissive hypercapnea. However, low-tidal volume ventilation has been recognized to decrease recruited lung volume, a phenomenon that persists despite the aggressive positive end-expiratory pressure (PEEP) strategy employed in ARDSNet studies. Atelectasis associated with low-tidal volume ventilation is relieved through the use of so-called sigh breaths, higher levels of PEEP or recruitment maneuverers. Further, the proportion of lung remaining in the derecruited state may contribute to the morbidity and mortality associated with ARDS. In adults, several strategies have been utilized to recruit the lung: sustained inflation (SI) and the maximal recruitment strategy. The so-called open lung approach (OLA) includes an SI followed by the setting of PEEP to the measured lower inflection point of the PV curve. An alternative approach to setting PEEP is a decremental PEEP titration, which includes the sequential lowering of PEEP until a predetermined decrement in PaO2 or SaO2 occurs.

The impact of lung recruitment in the long-term course of ARDS is not yet clear. It is clear that lung recruitment is most effective earlier in the course of ARDS. Grasso et al demonstrated that patients who received a recruitment maneuver on day 1±0.3 of ARDS could be recruited, versus patients recruited on day 7±1. Similarly, Gattinoni et al7 and Crotti et al found limited recruitment in patients who were well along in the course of ARDS. Borges et al, Tugrul et al, and Girgis et al all recruited patients early in the course of ARDS, and each found marked lung recruitment, on average, in all the patients studied. Each of these studied demonstrated an ability to improve oxygen saturations and (sometimes studied) end-expiratory lung volume. While no study has examined the effect of this change on morbidity or mortality, in children hypoxemia is known to be a common cause of morbidity. Importantly in children, treatment of hypoxia often drives escalating ventilator settings, the use of high frequency oscillatory ventilation (HFOV) or the use of extra-corporeal membrane oxygenation (ECMO). Early recruitment and proper titration of PEEP in children with ARDS may prevent the need for escalation of care towards these more invasive, and risk-imposing therapies.

Electrical Impedance Tomography (EIT) Barber and Brown introduced electrical impedance tomography to the medical community in the early 1980s. From there a wide spectrum of applications in medicine ranging from gastric emptying, brain function, breast imaging, to lung function have been explored. It is our belief that the most valuable benefit of EIT is in the monitoring of regional lung function in critically ill patients. Early EIT devices fell susceptible to poor sensitivity and signal interference in the clinical setting. After years and a renewed interest from a few commercial companies interested in ventilation technology, many of these shortcomings have been resolved. As with any new modality, EIT and its clinical utility and application need to be methodically explored; therefore we propose this IRB protocol to take us a step closer on this journey to develop a clinically useful tool.

Electrical impedance tomography capitalizes on changes in electrical impendence between air-filled versus tissue or fluid-filled spaces in order to characterize and quantify regional distribution of lung volume at the bedside. This technology has been validated in animal and human studies. The technology utilizes a series of 16 electrodes placed across the patient's chest. As small currents, which are undetectable to the subject, are passed between the electrodes, impedance is measured between and amongst the series. Through a complex interrogation and manipulation of these impedance values, a two-dimensional image is formed, and has been shown to correlate with clinical and radiographic changes in patients. The ability to estimate lung volume and regional distribution of gas non-invasively and in real time may give us insight as to what mode of ventilation or setting is more effective in optimizing positive pressure ventilation.

ELIGIBILITY:
Inclusion Criteria:

1. All intubated and mechanically ventilated patients will be screened for the following inclusion criteria: 2. Age: Age 2 to 35 years 3. Arterial line 4. Have ARDS based on the following definition:

a. The Berlin definition of ARDS36 i. Blood gas criteria:

1. Mild: PaO2/FiO2 ratio of 201-300,
2. Moderate: PaO2/FIO2 ratio of 101-200
3. Severe: PaO2/FIO2 ratio of < 100 ii. Acute onset (within 1 week) of bilateral (patchy, diffuse, or homogeneous) infiltrates consistent with pulmonary edema on chest radiograph, and iii. No evidence of left atrial hypertension

5. Conventional lung protective mechanical ventilation Chest radiograph within the first 12h after the study recruitment

Exclusion Criteria:

1. Meets the above criteria for ARDS for > 72 hours
2. < 2 years of age or chest circumference < 55 cm.
3. Clinically recognized airways disease (e.g. anatomic or reactive airway disease by history, treatment or flow graphics)
4. Uncuffed endotracheal tube in place
5. Airleak
6. Congenital heart disease
7. Hemodynamically significant heart disease
8. Congenital diaphragmatic hernia
9. Pulmonary fibrosis
10. Restrictive lung disease (other than ARDS)
11. Cystic fibrosis
12. Significant pulmonary hypertension requiring treatment (eg iNO, sildenafil, flolan)
13. Severe brain injury with no intracranial pressure monitor or external ventricular drain in place
14. Extra-corporeal life support
15. Patients with unstable spinal injuries or diseases
16. Body mass index > 50
17. Active implant such as pacemaker, ICD, or diaphragm pacer
18. Skin integrity issues in the area that the belt / electrodes will be placed, such as ulcers or open wounds
19. Dressings or chest tubes that prohibit the placement of electrodes in the proper plain.
20. Open chest
21. Flail chest within the regional plain of the belt / electrodes
22. If the medical team feels that the patient is not appropriate to enroll in the study based on medical, social or emotional concerns
23. If the patient is too unstable to position the belt / electrodes and/or transition to the Draeger ventilator

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 0 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Safety - measured by Barotrauma | 3 days
Safety - measured by Gas Exchange | 3 days

CONTACTS AND LOCATIONS:
Locations (1):
- Boston Children's Hospital, Boston, Massachusetts, United States